CLINICAL TRIAL: NCT05780112
Title: Evaluation of The Effectiveness of The Breathing Exercise On The Nausea, Vomiting And Quality of Life In The Early Pregnancy Period: A Single-Blind Randomized Controlled Trial
Brief Title: The Effectiveness of The Breathing Exercise On The Nausea, Vomiting And Breathing Exercise In Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Tülay AYTEKİN AYDIN, Women's Health and Diseases Nurse, Inonu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019/6-28
Record Dates: First submitted 2022-01-05; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy
Keywords: Breathing Exercise; Nausea and Vomiting; Nursing; Pregnancy; Quality of Life
MeSH Terms: conditions — Nausea; Vomiting | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The pregnant women did the breathing exercise in accordance with the 'Practical Guideline on Breathing Exercise for Reducing Nausea and Vomiting in the Pregnant Women'. The breathing exercise training took on average 15-20 minutes for each pregnant woman. After the training, the pregnant women were asked to do the breathing exercise properly and effectively in accordance with the guideline for a minimum of five minutes at least twice a day for four weeks.
  * Refresher training was given to the pregnant women through phone calls at the end of the first and third weeks and home visits at the end of the second week, and in each of these interviews, the pregnant women's breathing exercise practices were followed and the NVPI was applied to the pregnant women.
  * At the end of the research, in other words, at the end of the fourth week, the NVPI and SF-36 were applied once again to the pregnant women in the maternity polyclinic, and hence, the follow-up process came to an end.
  Interventions: Other: breathing exercise
- control group (No Intervention): At the beginning of the research (pretest phase), without giving information about the breathing exercise practice to the pregnant women and making them practice the exercise, the researcher only asked pregnant women in the control group to fill in the Personal Information Form and applied the NVPI and SF-36 to the pregnant women.
  * The pregnant women were called by phone at the end of the first and third weeks and their homes were visited at the end of the second week, and in each interview, information about their health status was received from them and the NVPI was applied to them.
  * At the end of the research (post-test phase), in other words, at the end of the fourth week, the NVPI and SF-36 were applied once again to the pregnant women in the maternity polyclinic.

INTERVENTIONS:
Other: breathing exercise — * Place one hand on your chest and the other on your stomach.
  * Slowly take a deep breath through the nose.
  * During inhalation, your hand on your stomach should rise upwards as the air fills the lungs. If it is under your hand on the chest, there should not be much movement.
  * Hold your breath and stretch your muscles in a second or two.
  * Take air through your nose with your mouth closed and exhale slowly through your mouth by pursing your lips like a whistle.
  * Set the time you use when exhaling air to be twice the time you use when exhaling.
  * As you exhale, focus on the inward movement of your abdominal hand.
  Arms: Experimental group

SUMMARY:
Aim: This study aimed to investigate the effectiveness of the breathing exercise on pregnancy-related nausea and vomiting and the quality of life in the early pregnancy period.

Background: Nausea and vomiting during pregnancy is a condition that can negatively affect the quality of life and the course of pregnancy in pregnant women. Nausea and vomiting during pregnancy with breathing exercises and can positively affect the quality of life women.

Methods: This study is a single-blind randomised controlled trial. The sample consisted of 104 pregnant women. The Personal Information Form, the Nausea and Vomiting in Pregnancy Instrument and the 36-Item Short-Form Health Survey were used to collected the data.

DETAILED DESCRIPTION:
2.1. Study design, sampling and recruitment strategies This research was conducted as a randomized controlled experimental study with the pretest-posttest design. The research was carried out in the maternity polyclinic of a public hospital affiliated with the Health Directorate of Elazığ Province in eastern Turkey in June 2019 - May 2020. A total of 104 pregnant women took part in the research (52 pregnant women in the experimental group and 52 pregnant women in the control group). In the calculation of the sample size, the power analysis was utilized. Considering that the effect of the breathing exercise on nausea and vomiting and the quality of life in the early pregnancy period will increase the mean of the Nausea and Vomiting in Pregnancy Instrument scores eight points after the breathing exercise, the number of participants for each group was calculated as 52 pregnant women at α=0.05 significance level and with 80% power [1-β (power)=0.80].

In the research, the inclusion criteria were designated as follows: a) Having the ability to communicate, b) Being aged 15-49 years, c) Being in the 12th or an earlier week of pregnancy with a living fetus, d) Not having fetal congenital malformation, e) Not having systemic diseases (gastrointestinal system, audiovestibular, endocrine, infection, and psychological diseases) which are likely to lead to nausea and vomiting other than pregnancy-related nausea and vomiting, f) never using a medication against nausea and vomiting before.

Under the research, the following were identified as the exclusion criteria: a) Having a multiple pregnancy, b) Having fetal congenital malformation, c) Having systemic diseases that are likely to lead to nausea and vomiting, d) Using medication against nausea and vomiting, e) Having the risk of miscarriage, f) Having speech disorder.

2.2. Instruments In the collection of research data, the Personal Information Form, the Nausea and Vomiting in Pregnancy Instrument, and the 36-Item Short-Form Health Survey were used. The research data were gathered by the researcher using the face-to-face interview technique.

2.2.1. Personal Information Form In the Personal Information Form which was prepared by the researcher as per the literature review (Şahan, 2012; Acog Practıce Bulletın, 2018; Köken et. al., 2009; Aksu, & Şirin 2007), seven questions addressed the pregnant women's socio-demographic characteristics (age, education, employment status, income level, body mass index-BMI) and ten questions pertained to the pregnancy (the number of previous pregnancies, whether the pregnancy was unwanted or not, the number of nausea and vomiting per day, and so on.), and hence, the form contained 17 questions in total.

2.2.2. Nausea and Vomiting in Pregnancy Instrument (NVPI) The Nausea and Vomiting in Pregnancy Instrument was developed by Swallow et al. (2002) for evaluating nausea and vomiting during pregnancy 'within the last week'. The NVPI was used after the time frame was re-configured as 'the week in which the pregnant woman had nausea and vomiting most frequently'. The NVPI is comprised of three questions that addressed the frequency of nausea, retching, and vomiting for one week. Each question was scored on the basis of a 6-point Likert scale. The scores to be obtained from each NVPI question ranged from 0 to 5 points, and the minimum and maximum scores to be obtained from the NVPI were respectively 0 and 15 points. There is no cut-off point for the NVPI. The increase in the NVPI scores demonstrates that the severity of nausea and vomiting rose (49, 79). This measurement tool was used for evaluating the severity of nausea, retching, and vomiting through the weekly follow-ups of the individuals.

2.2.3. 36-Item Short-Form Health Survey (SF-36) The SF-36 was developed by Ware (1992). The validity and reliability test for the SF-36 was performed in Turkey by Pınar (1995), and it was asserted that the SF-36 was applicable to chronic diseases (Acaray, & Pınar, 2004; Tel, 2009). As the name suggests, the SF-36 is composed of 36 questions and eight sub-scales (physical functioning, role physical, bodily pain, general health perceptions, vitality, social functioning, role emotional, and mental health) (Ware, & Sherbourne, 1992; Koçyiğit et. al., 1999). Just as the SF-36 and its eight sub-scales are evaluated separately, the SF-36 can also be evaluated under two main dimensions, namely, physical dimension and mental dimension. The physical dimension covers the domains of physical functioning, role physical, bodily pain, general health perceptions, and vitality while the mental dimension includes the domains of social functioning, role emotional, mental health, general health perceptions, and vitality. For the physical and mental dimensions, the mid-range value was set as 50 points, and the scores above and below 50 points are successively categorized as being above and below the mid-range. The questions are scored through a Likert scale and cover the last four weeks (Acaray, & Pınar, 2004; Tel, 2009).

The SF-36 is evaluated differently for each sub-scale. The fourth and fifth questions of the SF-36 are dichotomous questions evaluated and scored as either yes or no whilst the rest of the questions are scored as per 3-point, 5-point, and 6-point Likert scales. The items 1, 6, 7, 8, 9d, 9e, 9h, 10b, and 10d under the SF-36 are reverse-scored. The sub-scales evaluate the state of health based on scores that range from 0 to 100 points. A score of 0 represents 'bad health' whereas a score of 100 is denoted as 'good health' (Ware, & Sherbourne, 1992; Koçyiğit et. al., 1999). Cronbach's Alpha coefficient was calculated as 0.93 for the SF-36 (Koçyiğit et. al., 1999). Under this research, Cronbach's Alpha coefficient was identified as 0.86 for the SF-36.

2.3. Randomization The research was carried out with the pregnant women who had nausea and vomiting, applied to the hospital (polyclinic) and agreed to participate in the research. Information about the research procedure was given to the participant pregnant women, and all participants were required to fill in the informed consent forms before the randomization process. Then, they were randomly assigned to the experimental or control groups. The simple random sampling, a probability sampling method, was used in the selection of the participant pregnant women, and the random sampling was continued until the sample size reached the designated number of participants. The randomization was performed through the generation of random numbers via MedCalc 18.2.1 software. All participant pregnant women were blinded to the randomization process. However, it was not possible to blind the researcher to the breathing exercise due to the nature of this intervention (Figure 1).

2.4. Research Process Before conducting the research, the researcher contacted the physician responsible for the unit and the nurses working for the unit and introduced herself and the study. Next, the pregnant women satisfying the inclusion criteria which were designated for the research were identified and randomly assigned to the experimental and control groups. The 'experimental group' was made up of the pregnant women who did breathing exercises whereas the 'control group' was composed of the pregnant women who did no breathing exercise. In the interview held with the pregnant women in the maternity polyclinic, the researcher informed them about the study and asked them to give their informed consent in written format and verbally.

Experimental Group:

* At the beginning of the research (pretest phase), information about how the research would be conducted was given to each participant pregnant woman in the experimental group, and the pregnant women in the experimental group were informed that they were free to leave the research any time they wanted and they were invited to take part in the research. Next, the pregnant women in the experimental group were asked to fill in the Personal Information Form, and subsequently, the NVPI and SF-36 were applied to them, and afterward, the training about the application of the breathing exercise was offered to them.
* The pregnant women did the breathing exercise in accordance with the 'Practical Guideline on Breathing Exercise for Reducing Nausea and Vomiting in the Pregnant Women' which was prepared by the researcher in light of the relevant literature (Bustos, 2017; Aşçı, & Özer, 2011; Aksu, & Şirin 2007; Song et. al., 2013; Ölçer, & Oskay 2015). This guideline was developed as per the expert opinions and included the application steps of the breathing exercise. First, by doing the breathing exercise in accordance with the guideline, the researcher provided the pregnant women with a show of how to do the breathing exercise, and then, asked them to practice this exercise. The breathing exercise training took on average 15-20 minutes for each pregnant woman. After the training, a copy of the 'Practical Guideline on Breathing Exercise for Reducing Nausea and Vomiting in the Pregnant Women' was given to all pregnant women, and the pregnant women were asked to do the breathing exercise properly and effectively in accordance with the guideline for a minimum of five minutes at least twice a day for four weeks.
* Refresher training was given to the pregnant women through phone calls at the end of the first and third weeks and home visits at the end of the second week, and in each of these interviews, the pregnant women's breathing exercise practices were followed and the NVPI was applied to the pregnant women.
* At the end of the research (post-test phase), in other words, at the end of the fourth week, the NVPI and SF-36 were applied once again to the pregnant women in the maternity polyclinic, and hence, the follow-up process came to an end.

Control Group:

* The pregnant women in the control group were informed that they would be followed each week for nausea and vomiting and were free to leave the research any time they wanted, and they were invited to participate in the research.
* At the beginning of the research (pretest phase), without giving information about the breathing exercise practice to the pregnant women and making them practice the exercise, the researcher only asked pregnant women in the control group to fill in the Personal Information Form and applied the NVPI and SF-36 to the pregnant women.
* The pregnant women were called by phone at the end of the first and third weeks and their homes were visited at the end of the second week, and in each interview, information about their health status was received from them and the NVPI was applied to them.
* At the end of the research (post-test phase), in other words, at the end of the fourth week, the NVPI and SF-36 were applied once again to the pregnant women in the maternity polyclinic.
* At the end of the study, on a voluntary basis, the pregnant women in the control group were informed about the deep breathing exercise, and the 'Practical Guideline on Breathing Exercise for Reducing Nausea and Vomiting in the Pregnant Women' was given to them. The pregnant women were advised to do this breathing exercise properly and effectively when they felt nausea, and accordingly, the follow-up procedure was finalized for them.

2.5. Data analysis The statistical analysis of the research data was performed with the IBM SPSS 22.0 (Statistical Package for the Social Science). In the analysis, the mean±standard deviation, and median (min-max) were used for evaluating the numerical data whilst the frequency and number (percentage) statistics were utilized for evaluating the nominal (demographic) data. Whether the research data had normal distribution was checked with the Shapiro-Wilk test. The student t-test was employed in the inter-group comparisons of the normally distributed variables while the Mann-Whitney U test was used for the inter-group comparisons of the variables with non-normal distribution. In the two dependent group comparisons of the normally distributed variables, the paired t-test was utilized. The relationship between the categorical variables was analyzed using the Pearson chi-squared test. The reliability of the measurement tools was evaluated with Cronbach's Alpha coefficient. The statistical significance was identified if the P-value was lower than 0.05 (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to communicate,
* Being aged 15-49 years,
* Being in the 12th or an earlier week of pregnancy with a living fetus,
* Not having fetal congenital malformation,
* Not having systemic diseases (gastrointestinal system, audiovestibular, endocrine, infection, and psychological diseases) which are likely to lead to nausea and vomiting other than pregnancy-related nausea and vomiting,
* never using a medication against nausea and vomiting before.

Exclusion Criteria:

* Having a multiple pregnancy,
* Having fetal congenital malformation,
* Having systemic diseases that are likely to lead to nausea and vomiting,
* Using medication against nausea and vomiting,
* Having the risk of miscarriage,
* Having speech disorder.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — pregnant women
Enrollment: 104 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Nausea and Vomiting in Pregnancy Instrument (NVPI) | Change from Nausea and Vomiting in Pregnancy Instrument at 4 weeks
  The Nausea and Vomiting in Pregnancy Instrument was developed by Swallow et al. (2002) for evaluating nausea and vomiting during pregnancy 'within the last week'. The NVPI was used after the time frame was re-configured as 'the week in which the pregnant woman had nausea and vomiting most frequently'. The NVPI is comprised of three questions that addressed the frequency of nausea, retching, and vomiting for one week. Each question was scored on the basis of a 6-point Likert scale. The scores to be obtained from each NVPI question ranged from 0 to 5 points, and the minimum and maximum scores to be obtained from the NVPI were respectively 0 and 15 points. There is no cut-off point for the NVPI. The increase in the NVPI scores demonstrates that the severity of nausea and vomiting rose
36-Item Short-Form Health Survey | Change from 36-Item Short-Form Health Survey Instrument at 4 weeks
  SF-36 is composed of 36 questions and eight sub-scales (physical functioning, role physical, bodily pain, general health perceptions, vitality, social functioning, role emotional, and mental health). ). Just as the SF-36 and its eight sub-scales are evaluated separately, the SF-36 can also be evaluated under two main dimensions, namely, physical dimension and mental dimension. The physical dimension covers the domains of physical functioning, role physical, bodily pain, general health perceptions, and vitality while the mental dimension includes the domains of social functioning, role emotional, mental health, general health perceptions, and vitality. For the physical and mental dimensions, the mid-range value was set as 50 points, and the scores above and below 50 points are successively categorized as being above and below the mid-range.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided